CLINICAL TRIAL: NCT05060913
Title: Upshots of 5% Emla Cream Versus 20% Benzocaine on Pre-Injection Analgesia.
Brief Title: Emla Cream Versus Benzocaine on Analgesia
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Shaharyar Hamid, Dr. Shaharyar Hamid, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ShHamid2190
Record Dates: First submitted 2021-09-18; First posted 2021-09-29 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Effect of Drug
MeSH Terms: interventions — Lidocaine, Prilocaine Drug Combination; Lidocaine; Prilocaine; Benzocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 5% EMLA Cream (Experimental): EMLA cream will be applied over buccal mucosa of one side for 1.5 minutes of Maxillary of Mandibular anterior teeth.
  Interventions: Drug: EMLA Cream
- 20% Benzocaine gel (Active Comparator): Benzocaine gel will be applied over buccal mucosa on another side for 1.5 minutes of Maxillary of Mandibular anterior teeth.
  Interventions: Drug: Benzocaine Gel

INTERVENTIONS:
Drug: EMLA Cream — Effect of 5% Emla cream on pricking pain measured on VAS scale.
  Other Names: 2.5% Lidocaine and 2.5% Prilocaine
  Arms: 5% EMLA Cream
Drug: Benzocaine Gel — Effect of 20% Benzocaine gel on pricking pain measured on VAS scale.
  Other Names: 20% Benzocaine
  Arms: 20% Benzocaine gel

SUMMARY:
EMLA is proven to be better in achieving pain control as topical anesthesia than benzocaine at palatal mucosa. So this research is done to compare its effectiveness at buccal mucosa.

Methods:

A total number of 70 patients attending DOW ojha hospital, fulfilling inclusion criteria and undergoing extraction of bilateral teeth will be included in this study. Approval of data collection will be sought from the Institutional ethical review board ¬(IERB) of Dow university of health sciences (DUHS) for this study. the participants will be briefed about the nature and purpose of the study including visual analogue scale (VAS). They will be ensured that their information will be used for the study purpose only. Informed consent from the participants will be obtained. Complete history from patients will be taken. The sites will be divided into condition A- 5% EMLA and Condition B - 20% Benzocaine Gel. After marking injection sites, principal investigator will leave the room and the consultant will apply 5% EMLA gel at experimental area and 20% Benzocaine gel at control area. After pre-treatment with topical anesthesia the consultant will administer local anesthesia to both sides. Then Principal investigator will be signaled into the room and patient will be assessed though visual analogue scale by him and will be confirmed by supervisor.

DETAILED DESCRIPTION:
The concept of dental pain is a true fear for many people. In dentistry, management of pain and anxiety has evolved through behavior modification and oral and intravenous sedatives. Whereas local anesthesia is known as the backbone of the profession. Over the years, methods have been introduced to reduce the pricking pain of local anesthesia injection. There are so many factors which help reduce the pain caused by local anesthesia injection such as warming the local anesthetic agent, specific size of needle gauge, a certain type of anesthetic solution and topical anesthetics. Topical anesthetics are used at insertion sites before injections to reduces the slight discomfort with insertion of the needle. [1,2,3] OneaofatheaTopicalaanesthetics widelyaused for dental proceduresaincludesaBenzocaine.[4] Benzocaine is anaFDA-approved drugawhichaisaavailable in various forms and concentrations. In the 20% concentration, benzocaineagel is the most commonly used topical anesthetic in dentistry, withaanaonsetatimeaofa30asecondsaandadurationaofa5-15aminutes. EMLA is a eutectic mixture of the two local anesthetics, prilocaine and lidocaine which melt at lower temperatures than any of its components, permitting higher concentrations of anesthetics for use.[5] It is used to reduce the pain associated with venous cannulation.

Past studies have reported the pharmacologic and the psychological effects on pain control by benzocaine and Eutectic mixture of local anesthetics (EMLA). However, there is no valuable data on the effect of the simultaneous use 5% EMLA and 20% Benzocaineaonapainaperceptionaduring injectionainaoralamucosaainapopulationaof Karachi. The presentastudyawasadesignedato evaluate the effect of topical application of 5% EMLAaand 20% Benzocaine in an adult population in reducing pain of injection of the local anesthetic agent.

Methods:

A total number of 70 patients attending DOW ojha hospital, fulfilling inclusion criteria and undergoing extraction of bilateral teeth will be included in this study. Approval of data collection will be sought from the Institutional ethical review board ¬(IERB) of Dow university of health sciences (DUHS) for this study. the participants will be briefed about the nature and purpose of the study including visual analogue scale (VAS). They will be ensured that their information will be used for the study purpose only. Informed consent from the participants will be obtained. Complete history from patients will be taken. The sites will be divided into condition A- 5% EMLA and Condition B - 20% Benzocaine Gel. After marking injection sites, principal investigator will leave the room and the consultant will apply 5% EMLA gel at experimental area and 20% Benzocaine gel at control area. After pre-treatment with topical anesthesia the consultant will administer local anesthesia to both sides. Then Principal investigator will be signaled into the room and patient will be assessed though visual analogue scale by him and will be confirmed by supervisor.

ELIGIBILITY:
Inclusion Criteria:

1. Patients indicated for bilateral extraction and requiring local anesthesia technique.
2. Patients in the age group of 18 to 35 years.
3. Patients willing to take part in study.

Exclusion Criteria:

1. Patients not willing to participate in the study
2. Patients presenting with local inflammation / tenderness at site of injection
3. Patients who are allergic to local anesthesia
4. Patients on antidepressant or anti-psychotic drugs
5. Patient with history of any medical condition.
6. Patient with history of methemoglobinemia

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2021-11-17 (Actual); Primary Completion 2022-03-02 (Actual); Study Completion 2022-03-04 (Actual)

PRIMARY OUTCOMES:
Achievement of local anesthesia | Reading on VAS will be taken after applying EMLA cream for 1.5 minutes.
  local anesthesia will be assessed with the help of Visual Analog Scale. VAS score must be '0' while pricking injection for applying Local anesthesia.
Achievement of local anesthesia | Reading on VAS will be taken after applying Benzocaine gel for 1.5 minutes.
  local anesthesia will be assessed with the help of Visual Analog Scale. VAS score must be '0' while pricking injection for applying Local anesthesia.

CONTACTS AND LOCATIONS:
Overall Officials: Shaharyar hamid, Principal Investigator — Dow University of Health Sciences
Locations (1):
- Dr. Ishrat-ul-Ebad institute of oral health sciences, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No